CLINICAL TRIAL: NCT03013049
Title: A Comparative Study Between Autologous Non Cultured Epidermal Cell Suspension Versus Combination of Autologous Non Cultured Epidermal Cell Suspension and Non Cultured Dermal Cell Suspension in Stable Vitiligo
Brief Title: A Novel Surgical Method in the Treatment of Unstable Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Davinder Parsad, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2016/2675
Record Dates: First submitted 2016-12-27; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non cultured epidermal cell suspension (Active Comparator): In 20 patients who have stable vitiligo with the duration of stability more than 3 months, non cultured epidermal cell suspension will be done. Patients will be divided into 2 subgroups of 10 patients each of stability duration of 3-6 months and more than 1 year respectively and non cultured epidermal cell suspension will be done.
  Interventions: Procedure: Non cultured epidermal cell suspension
- Non cultured dermal cell suspension (Experimental): In 20 patients who have stable vitiligo with the duration of stability more than 3 months, combination of non cultured epidermal cell suspension and non cultured dermal cell suspension will be done. Patients will be divided into 2 subgroups of 10 patients each of stability duration of 3-6 months and more than 1 year respectively and combination of non cultured epidermal cell suspension and non cultured dermal cell suspension will be done.
  Interventions: Procedure: Non cultured epidermal cell suspension; Procedure: Non cultured dermal cell suspension

INTERVENTIONS:
Procedure: Non cultured epidermal cell suspension — Non cultured epidermal cell suspension Split thickness skin specimen will be transferred under aseptic conditions to a container with normal salineand transferred to laboratory. There, the skin graft will be transferred to Trypsin-EDTA solution (0.25% trypsin and 0.02% EDTA) in a Petri dish and incubated overnight at 4°C in 5% CO2 to separate the epidermis from the dermis.Afterwards, the Trypsin-EDTA solution will be removed and PBS will be added and pipetted well so as to separate the cells from the tissue.The suspension will be centrifuged at 1000 rpm for 5 minutes.The supernatant will then be discarded and Phosphate buffer saline is added to make suspension of non-cultured epidermal cells.
Procedure: Non cultured dermal cell suspension — Non-cultured Dermal Cell Suspension Skin punch will be collected in phosphate buffer saline (PBS) with antibiotics (penicillin and streptomycin). The epidermis will be cut off from dermis carefully using a surgical blade (Epidermal part will be used for the epidermal cell suspension). Dermis will be then cut into small pieces and incubated in collagenase (1mg/ml) overnight at room temperature. Next day content will be diluted with PBS and centrifuged at 1000rpm for 5 minutes. Pellet will be washed three times with PBS to remove collagenase activity. Phosphate buffer saline is added to make suspension of non-cultured dermal cells and will be used for the autologous transplantation.
  Arms: Non cultured dermal cell suspension

SUMMARY:
Vitiligo is a complex disease causing a selective, often progressive, loss of functioning melanocytes from epidermal basal layer resulting in white patches on the skin and occasionally mucosae. Worldwide prevalence of vitiligo is around 1% whereas in India it is around 3-4% ranging from 0.46% to 8.8%.

Etiopathogenesis of vitiligo is multifactorial consisting of genetic, immunological and environmental factors. Environmental and genetic factors act in concert to destroy melanocytes. Reactive oxygen species (ROS) play important roles in vitiligo pathology,but the autoimmune pathogenesis has been proposed as one of the main causes of vitiligo.

Surgical methods, mainly transplantation of non cultured epidermal cell suspension are effective treatment for stable vitiligo. Transplantation of autologous noncultured epidermal cell suspension and non-cultured dermal cell suspension in combination (a mode of cellular grafting technique) is a novel surgical method for the treatment of vitiligo. Cytotoxic CD8+ ( cluster of differentiation 8+) cells in vitiligo perilesions may dictate the fate of transplantation, and strategies against CD8+ T cell activation might be beneficial for patients undergoing melanocyte transplantation. Mesenchymal cells could inhibit T cell proliferation and induce T cell apoptosis. Bartsch first identified and characterized dermal mesenchymal cells (DMCs). They have a multi-lineage differentiation potential into adipocytes, osteocytes and chondrocytes.Vitiligo patients' autologous melanocytes transplantation efficiency may be predicted by perilesional skin-homing CD8+ T cell activities, and the immunoregulatory DMCs might be used as auxiliary agent to improve the efficacy.

This pilot study is planned to compare transplantation of autologous noncultured epidermal cell suspension v/s its combination with non-cultured dermal cell suspension as a novel method in vitiligo surgery in stability of vitiligo with regards to extent of repigmentation, color matching of repigmented area, patient satisfaction and adverse events if any. This is the first study using transplantation of autologous noncultured epidermal cell suspension and non-cultured dermal cell suspension in combination as a new modality in vitiligo surgery.

DETAILED DESCRIPTION:
Vitiligo, the most common depigmenting disorder is an 'idiopathic', acquired pigmentary disorder caused by the loss of functional melanocytes from the epidermis. The course of the disease is unpredictable but is often progressive with phases of stabilized depigmentation. It usually begins during childhood or young adulthood. Approximately one third to one half of the patients develops the disease before the age of 20 years. The presence of vitiligo on exposed areas of body leads to social embarrassment, psychological turmoil, and cosmetic disfigurement in those affected.

Its prevalence is 1%, ranging from 0.1 to > 8.8% in different countries of the globe. Both sexes are equally affected although the greater number of reports among females is probably due to the greater social consequences to women and girls affected by this condition.

Treatment options A number of therapeutic options for vitiligo are available but there is still a need for a treatment that is promptly effective. There is no curative treatment for this condition. Management of vitiligo is a real challenge for a dermatologist.

Medical therapies:

Corticosteroids (Topical, intralesional and systemic), Oral mini pulse, PUVA (topical and systemic), NBUVB, calcipotriol and tacrolimus are used most widely. Some of the less commonly used medical modalities include phenylalanine, khellin, topical minoxidil, levamisole and melagenina. Recently oral minocycline was shown to be effective in treating vitiligo.

Most of these therapies aim to restore melanocyte function by their anti-inflammatory or immunomodulatory action and by preventing melanocyte auto destruction so that normal skin appearance and function is restored.

Surgical therapies:

All patients with vitiligo should be initially treated with medical methods. Surgical methods are important solutions for stable vitiligo refractory to medical treatment. High repigmentation rates are obtained with all procedures so far described in most anatomic locations, but they are of little help for acral areas and bony prominences. Unilateral vitiligo is the clinical form with the best response to grafting and transplant methods, and a good proportion of patients with stable bilateral disease also respond adequately. Nevertheless, appropriate patient selection is important to achieve maximal results.However none of the surgical modalities developed so far is uniformly effective in all patients and body sites and there is need for constant research and innovations for better surgical therapeutic options for vitiligo.

Aims of various surgical procedures:

A) Camouflage Tattooing: Introduction of artificial pigments into the lesions for permanent camouflage.

B) Excision: Removal of the depigmented areas, e.g. excision with primary closure and covering with thin Thiersch's graft.

C) Melanocyte transplantation: commonly used methods of autologous transplant of melanocytes are

Tissue grafts:

1. Thin and ultra-thin split thickness grafts (STSG)
2. Suction blister epidermal grafts(SBEG)
3. Mini punch grafts (MPG)
4. Hair follicular grafts (HFG)

   Cellular grafts:
5. Noncultured epidermal cell suspension (NCES)
6. Cultured "pure" melanocytes (CM)
7. Cultured epithelial grafts (CE)
8. Autologous noncultured extracted hair follicle outer root sheath cell suspension also called follicular cell suspension (FCS) D) Therapeutically wounding the lesion to stimulate the melanocytes from the periphery and the black hair follicles to proliferate, migrate and re-pigment the lesion, e.g. therapeutic dermabrasion, laser ablation, cryosurgery (liquid nitrogen spraying), needling and local application of phenol or trichloroacetic acid.

Every method has its own advantages and disadvantages. As there are no specific data available from the prospective studies in this field, it is not easy to recommend which surgical approach to vitiligo offers the best result.

'Vitiligo global issues consensus conference, 2011' convened by Vitiligo European Task Force (VETF), concluded that assessment of 'overall' stability is inaccurate and unreliable, whereas individual lesion stability is more reliable, especially when used in the context of surgical intervention.

Methods and Size of Lesions:

Depending on the size of the treated area, the method may vary. Simple methods such as mini punch grafting and suction epidermal grafting are useful for small or medium sized lesions. On the contrary, for extensive depigmented defects, cellular transplants may be required.

Age:

Because of the invasive nature of surgical procedures, they are not recommended in children; nevertheless, highly motivated adolescents can be treated under sedation or general anesthesia. Also, it is not surprising to see patients beyond the age of 50 years who may be interested in surgical repigmentation.

Psychological Aspects:

Some patients with high emotional trauma because of depigmentation may seek advice for invasive procedures. However, a psychological evaluation may be needed to ascertain the real need for surgical treatment.

Photographic Record:

Illustrations are recommended to help in determining the percentage of improvement, quality of repigmentation and possible side effects.

Patient's Expectations:

Repigmentation is not always comparable with normally pigmented skin and the final results vary considerably from patient to patient. However, most individuals are pleased with the achieved results; minor imperfections are far less important than the noticeable repigmentation of vitiliginous skin, mainly in ethnic skin patients with a dark complexion; sometimes surgical repigmentation may look even better than what is observed in many patients after medical therapy.

Method and Donor Site:

Appropriate training with a specific method is an important prerequisite for surgical therapy. Donor site should be as hidden as possible and the gluteal region may be suitable for this purpose in most patients.

Success rates of different surgical options:

Among all procedures, suction blister epidermal grafts and thin and ultra-thin split-thickness grafts seem to be the most effective procedures, with overall success rates of 80.3% (CI 76.4-84.2%) and 77.9% (CI 72.2-83.6%) respectively. But, a recent randomized study directly comparing NCES and SBEG showed NCES is significantly better than SBEG. Among cellular grafts, all techniques seem to be equally effective with success rates of 61.1% (CI 56.1-66.1%), 63.6% (CI 57.2-70%), and 63.6% (CI 55.8-70.6%) for noncultured epidermal cell suspension, cultured melanocytes and cultured epidermis respectively. The mean repigmentation with noncultured extracted outer root sheath cell suspension is about 65.7%).

NONCULTURED EPIDERMAL CELL SUSPENSION The technique of noncultured epidermal suspension was pioneered by Gauthier et al. The suspension was prepared by incubating the donor skin obtained from the scalp in trypsin 0.25% for 18 hrs. The suspension was injected into blisters raised by cryotherapy. Eight out of the 12 patients treated had > 70% repigmentation at the vitiligo site. It was proposed that the presence of keratinocytes in the suspension supplies essential growth factors for melanocyte growth. They stated that this technique could emerge as simple and effective alternative to the costly cultured melanocyte transplantation technique.

NON-CULTURED DERMAL CELL SUSPENSION

Dermal mesenchymal cells were originally isolated from the dermis of juvenile and adult mice by Toma et al., afterwards, same group identified such a cell population in human skin. Georg Bartsch firstly identified and characterized dermal mesenchymal cells (DMCs). DMCs had multi-lineage differentiation potential into adipocytes, osteocytes and chondrocytes. The surface antigenic profile of DMCs was positive for CD90 but differs in regard to negativity for CD34.

Zhou et al investigated the factors determining the efficiency of autologous melanocyte transplantation of vitiligo patients by focusing on perilesional skin homing CD8+ T lymphocytes, and studied the potential effects of dermal mesenchymal cells (DMCs) on CD8+ T cell activities in vitro. The patients with high number of perilesional CD8+ T cells were associated with poor repigmentation rate and a significant lesser number of CD8+ T cells was infiltrating in patients with excellent or good re-pigmentation responses. Also, skin homing CD8+ T cells proliferation was significantly inhibited when co-culture with DMCs at 1:1 ratio as the percentage of proliferative CD8+ T cells dropped from 94.72% to 39.50% (p,0.05) after DMCs co-culture. In the co-culture system, DMCs significantly inhibited skin homing CD8+ T proliferation and induced those cells apoptosis. These data confirm that DMCs induces significant immunosuppressive abilities against skin homing CD8+ T lymphocytes and may help improve the efficacy of melanocytes transplantation. Non-cultured Dermal Cell Suspension (NDCS) is a novel method to increase the efficacy of non-cultured epidermal cell suspension (NCES).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinical diagnosis of focal, segmental or generalized vitiligo which has been stable for more than 3 months.

Exclusion Criteria:

1. Age less than 18 years
2. Pregnancy
3. Patient with actively spreading vitiligo
4. Appearance of new lesions
5. History of Koebnerisation
6. History of hypertrophic scars or keloidal tendency
7. Bleeding disorders
8. Patients with unrealistic expectation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
extent of repigmentation | 6 months
  Repigmentation will be assessed as follows -
  ≤25% Minimal repigmentation 26-50% Mild repigmentation 51-75% Moderate repigmentation 76-90% Marked repigmentation >90% Excellent repigmentation

SECONDARY OUTCOMES:
pattern of repigmentation | 6 months
  diffuse peri follicular migrating from the borders

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thakur V, Kumar S, Kumaran MS, Kaushik H, Srivastava N, Parsad D. Efficacy of Transplantation of Combination of Noncultured Dermal and Epidermal Cell Suspension vs Epidermal Cell Suspension Alone in Vitiligo: A Randomized Clinical Trial. JAMA Dermatol. 2019 Feb 1;155(2):204-210. doi: 10.1001/jamadermatol.2018.4919. PMID 30601885